Official Title: A Phase II Trial of Tildrakizumab for Prevention of Acute Graft-Versus-Host

Disease

NCT Number: NCT04112810

Date: December 13, 2022

Clinical Interventions template - Version: March 30, 2018

IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# Medical College of Wisconsin and Froedtert Hospital INTRODUCTION TO THE INFORMED CONSENT

| Name of Subject: |
|------------------|
| Name of Subject: |

IIT-Runaas-Tildrakizumab- A Phase II Trial of Tildrakizumab for Prevention of Acute Graft-Versus-Host Disease

Lyndsey Runaas, MD
Froedtert & Medical College of Wisconsin
Division of Hematology and Oncology
9200 W. Wisconsin Avenue
Milwaukee, WI 53226
414-805-6700

You are invited to take part in this research. You can decide whether to take part in this project or not. You are free to say yes or no. If there is anything that you do not understand, please ask questions.

# **Definitions**

**Allogenic HCT:** unrelated donor bone marrow transplant

**GVHD:** Graft versus Host Disease: a complication that can occur after an

allogeneic bone marrow transplant

HLA: human Leukocyte antigen. Proteins that help the body's immune system tell the

difference between its own cells and foreign, harmful substances

PFT: Pulmonary function test


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# **Purpose**

This project is being done to find out if giving Tildrakizumab in combination with standard GVHD prophylaxis; Tacrolimus and Methotrexate will help prevent acute and chronic GVHD.

### Length

1. You will be in this research project for about 12 months following your bone marrow transplant.

# **Procedures**

You will receive Tildrakizumab in combination with standard GVHD prophylaxis.

#### List of visits:

- Screening Visit
  - Total Number: 1
  - Total Time: approximately 2 to 4 hours
- Study drug Treatment Visits
  - Total Number: 5
  - Total Time: <u>approximately 1</u> hour each visit
- End of Treatment Visits
  - Total Number: 1
  - Total Time: approximately 2 to 4 hours

# Procedures that will occur at various visits:

# **Invasive Procedures**

 Drug administration, blood sample collection, and bone marrow/aspirate collection

#### **Non-invasive Procedures**

Full medical history exam, physical exam, pulmonary function tests

# Risks

This is a brief list of the most commonly seen side effects. The *full consent form* after this introduction contains a more complete list of potential research risks.

# Tildrakizumab and Standard GVHD Prophylaxis risks:

## Tildrakizumab:

- Hypersensitivity reactions: allergic reactions
- Respiratory: upper respiratory tract infections, pharyngitis
- Gastrointestinal: Nausea
- Hepatic: abnormal liver tests elevation
- Neurologic: headache, dizziness, lethargy (lack of energy)
- Cardiovascular: hypertension
- Insomnia-not able to sleep
- Dermatologic: skin rash, injection site erythema (reddening of the skin as a result of the injection)

### **Tacrolimus & Methotrexate:**

Discussed in C2


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# **Benefits**

We don't know if this project will help you. Your condition may get better but it could stay the same or even get worse.

# My Other Options

You do not have to join this project. Your other options may include:

- 1. Joining a different project
- 2. Routine care for this condition
- 3. Getting no treatment for this condition

If you have more questions about this project at any time, you can call Dr. Runaas at 414-805-6700.

If you have questions about your rights as a participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

#### CONSENT TO PARTICIPATE IN RESEARCH

#### A1. INTRODUCTION – WHY ARE WE ASKING YOU TO PARTICIPATE?

You are being invited to participate in this research because you have a type of cancer that will be treated with an allogenic HCT. Developing acute GVHD is a risk of this type of transplant. Because of your condition, you may be eligible for a research project using an investigational drug, Tildrakizumab, and standard GVHD prophylaxis to treat your disease.

A total of about 55 people are expected to participate in this research at the Medical College of Wisconsin/Froedtert Hospital.

The Director of the project is Lyndsey Runaas, MD in the Division of Hematology & Oncology. A research team works with Dr. Runaas. You can ask who these people are.

Sun Pharmaceuticals is providing support for this study.

#### A2. DO I HAVE TO PARTICIPATE?

You can decide whether to take part in this research or not. You are free to say yes or no. If you say no, your regular medical care will not change. Even if you join this project, you do not have to stay in it. You may stop at any time.

A research project is different from routine medical care in three ways: 1) there are extra risks that we will tell you about in this form; 2) you may have some extra medical tests and visits; 3) the research procedures, tests and visits follow a set plan that must be kept.

# A3. WHY IS THIS PROJECT BEING DONE?

In this study we want to find out if giving Tildrakizumab (100 mg) as a subcutaneous injection on Day -1 in combination with the standard GVHD prophylaxis; Tacrolimus and Methotrexate will help prevent acute and chronic GVHD. Tildrakizumab (100 mg) subcutaneous injection will also be given on Day +28, Day +112, Day +196 and Day +280 after your bone marrow transplant. We also want to find out whether the investigational drug combination is safe to use and whether it reduces the symptoms of acute and chronic GVHD.

Everyone in this study will receive the combination of Tildrakizumab and standard GVHD prophylaxis. This research and your samples will help us in creating controls and active drug levels for future research studies. The combination of Tildrakizumab and standard GVHD prophylaxis is still experimental and is not approved by the U.S. Food and Drug Administration.


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# **B1. WHAT WILL HAPPEN IF I PARTICIPATE?**

### **Treatment Schedule**

| | Days | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-<br>transpl<br>ant | -1 | 0 | +1 | +3 | +5 | +6 | +11 | +28 | +35 | +90 | +100 | +112 | +180 | +196 | +280 |
| Conditioning | Х | | | | | | | | | | | | | | | |
| Transplant | | | Χ | | | | | | | | | | | | | |
| Methotrexate | | | | Χ | Χ | | Χ | Χ | | | | | | | | |
| Tildrakizumab | | Χ | | | | | | | Χ | | | | X | | X | X |
| Tacrolimus | X | | | | Χ | | | | | | Taper* | X | X | Stop* | | |
| G-CSF | | | | | | Start^ | | | | | | | | | | |

<sup>\*</sup>If there is no evidence of GVHD

# Before the research starts (screening):

After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

# Screening procedures:

If the screening information shows that you meet the requirements, then you will complete the following:

- Medical History, which includes questions about your health, current medications.
- Physical Exam, which includes your height, weight
- Your performance status, which evaluates how you are able to carry on with your usual activities.
- Routine Blood tests (about 4 tablespoons)
- Pregnancy test if you are able to have children
- Infections disease markers
- HLA typing
- PFT: to test the function of your lungs
- Bone marrow biopsy and/or aspirate, to evaluate the extent of your disease. For this
  test, a sample of bone marrow cells is taken by a needle inserted into a bone in your
  body. If a bone marrow biopsy is needed, a small piece of bone and the attached bone
  marrow is removed. These tests may be done under local anesthesia.
- Research blood samples (approximately 4 teaspoons) to help understand the changes that are happening with your immune system to prevent GVHD

If the screening information shows that you cannot be in the research, the research doctor will discuss other options with you and/or refer you back to your regular doctor.


<sup>^</sup>G-CSF begins on day +5 after stem cell infusion and continues until engraftment is seen


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# Summary of Procedures: Day 0 to 365

# (See Table 1 for more detail)

- Physical Exam, which includes your weight
- Review of any side effects that you may be experiencing
- Routine Blood tests about 1 to 4 tablespoons at each timepoint listed on Table 1.
- Chimerism (engraftment analysis)
- PFT: to test the function of your lungs
- Bone marrow biopsy and/or aspirate, to evaluate the extent of your disease. For this
  test, a sample of bone marrow cells is taken by a needle inserted into a bone in your
  body. If a bone marrow biopsy is needed, a small piece of bone and the attached bone
  marrow is removed. These tests may be done under local anesthesia. Any time a bone
  marrow exam is done in the study, a sample will also be sent to a laboratory for research
  studies
- GVHD Assessments will be performed to determine if you are developing side effects as a result of the treatment you have been given. This assessment will be part of the physical exam.
- Research blood samples (approximately 32 teaspoons) to help understand the changes that are happening with your immune system to prevent GVHD
- Research stool samples to help understand the changes that are happening with your gut microbiome during study treatment
- Blood samples for pharmacokinetic labs and anti-drug antibody (ADA) testing (approximately 2 teaspoons) to help understand the way the drug is used and processed by your body
- Tildrakizumab subcutaneous injection: Day-1, Day+28, Day + 112, Day + 196, Day +280


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# Table 1

| Study Assessments | Baseline | Pre-<br>Trans<br>-plant | | Follow-up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Otady Assessments | Screening<br>Within 30<br>days prior<br>to infusion | Day -<br>1 | 28± 3<br>days | 56 +/-<br>7 days | 100<br>+/- 14<br>days | 112±<br>7 | 180+/<br>- 14<br>days | 196±<br>14 | 280±<br>14 | 12 month<br>post HCT (+/-<br>30 days) |
| Informed consent | X | | | | | | | | | |
| Tildrakizumab administration – 100 mg subcutaneously | | X | X | | | Х | | Х | X | |
| History, physical exam, weight, height | X | | Х | X | Χ | Х | X | Х | X | Х |
| HLA typing (donor and recipient) | X | | | | | | | | | |
| CBC with differential,<br>Comprehensive metabolic<br>panel | Х | | X | X | Х | Х | Х | Х | X | Х |
| Infectious disease markers^ | X | | | | | | | | | |
| LVEF | X | | | | | | | | | |
| DLCO and FEV1 | Х | | | | | | Х | | | X |
| Disease evaluation | Х | | | | Х | | | | | Х |
| Pregnancy test | X | | | | | | | | | |
| GVHD assessments | | | X | X | X | Χ | X | X | Χ | X |
| AE assessments | X | | X | Χ | X | Χ | X | X | Χ | |
| Chimerism | | | X | | | | | | | X |
| CMV NAAT peripheral blood | | | X | X | X | Χ | | | | |
| EBV PCR peripheral blood | | | Χ | Х | X | Χ | | | | |
| Immune reconstitution | | | X X X X | | | | | | | |
| Research blood and plasma | Х | Baseline (screening) and Days 7±3, 14±3, 21±3, 28±7, 60±14, 90±14, 196±30, 365±30 post-transplants and at the time of development of GVHD (if it occurs). | | | | | | | | |
| Research stool samples | | Days -1, 1±2, 7±2, 15±2, 21±2, until neutrophil engraftment with final stool sample collected after neutrophil engraftment. Will also be collected at the time of development of GVHD (if it occurs). | | | | | | | | |
| Pharmacokinetic labs and ADA testing | Х | Days 30±2, 60±7, and 90±14 | | | | | | | | |
| | | *For acute leukemia, CML, and MDS, this includes a bone marrow aspirate and biopsy and cytogenetics. ^CMV antibody, Hepatitis panel (HepA, HepB Sab, Hep B) | | | | | | | | |


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

#### **B2. HOW LONG WILL I BE IN THE PROJECT?**

You will be in this research project for about 12 months following your bone marrow transplant.

#### **B3. CAN I STOP BEING IN THE PROJECT?**

You are free to withdraw from the project at any time. If you leave, your regular medical care will not change. If you are thinking about leaving, please tell the research doctor.

- ⇒ The research doctor can tell you about the effects of stopping, and you and the research doctor can talk about what follow-up care would help you the most.
- ⇒ You might be asked to come back for one more visit to check your health.

The research doctor may take you out of this project at any time. This would happen if:

- They think it is in your best interest.
- You do not follow the project rules.
- The whole project is stopped.

If this happens, the research doctor will tell you.

#### **B4. ARE THERE ANY SPECIAL INSTRUCTIONS WHILE I AM IN THE PROJECT?**

- While you are participating in this study (during treatment), you can participate in other research studies as long as they are NOT GVHD prevention or treatment.
- You should also report to your doctor any changes in your health or side effects that you
  may be experiencing.
- You will be asked to receive all study-required treatments and complete all study-required procedures.

#### C1. WHAT HEALTH RISKS OR PROBLEMS CAN I EXPECT FROM THE PROJECT?

There are risks to taking part in any research project. There is a risk that you may get a drug combination that does not help your condition or may make it worse. There also may be problems (side effects) we do not know about yet, from the combination of Tildrakizumab and standard GVHD prophylaxis themselves, or how they combine with other drugs you are taking. If we learn about new important side effects, we will tell you.

We watch everyone in the project for problems (side effects). You need to tell the research doctor or a member of the research team immediately if you experience any problems, side effects, or changes in your health. If you have signs of fever or other new abnormal symptoms, call Dr. Runaas immediately at 414-805-6700. In an emergency, call 911.


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# C2. RISKS OF <u>TILDRAKIZUMAB IN COMBINATION WITH STANDARD GVHD</u> PROPHYLAXIS

The research drugs themselves may cause problems (side effects). Side effects may be mild or very serious. Some can last a long time or never go away.

The side effects that other people have experienced so far with the drug combination are:

# Tildrakizumab:

- Hypersensitivity reactions: allergic reactions
- Respiratory: upper respiratory tract infections, pharyngitis
- Gastrointestinal: Nausea
- Hepatic: abnormal liver tests elevation
- Neurologic: headache, dizziness, lethargy (lack of energy)
- Cardiovascular: hypertension
- Insomnia-not able to sleep
- Dermatologic: skin rash, injection site erythema (reddening of the skin as a result of the injection)

#### **Tacrolimus:**

- Cardiovascular: hypertension
- Neurologic: confusion, dizziness, insomnia, seizures, tremors, changes in how clearly one can think
- Gastrointestinal: nausea, vomiting
- Hematologic: microangiopathic hemolytic anemia (possible destruction of red blood cells), thrombocytopenia
- Endocrine and metabolic: hypomagnesemia (low blood level of magnesium), hypokalemia (low blood level of potassium), hypocalcemia (low blood level of calcium), hyperlipidemia (increase lipid level in blood)
- Miscellaneous: unwanted hair growth, changes in vision, liver problems, reversible renal insufficiency, infections and posttransplant lymphoproliferative disorders

#### Methotrexate:

- Neurologic: fever, dizziness, chills, undue fatigue
- Gastrointestinal: ulcerative stomatitis (painful swelling and sores inside the mouth), nausea, abdominal distress, diarrhea
- Hematologic: leucopenia (decreased number of white blood cells), anemia (decreased number of red blood cells)
- Miscellaneous: abnormal liver tests, kidney failure and pulmonary complications after transplantation

# C3. OTHER RISKS OF THIS RESEARCH PROJECT

Other procedures that are part of the research also involve some risks:


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# Blood Draws (for research blood and plasma, and pharmacokinetic labs)

Having your blood drawn can be uncomfortable and can sometimes cause a bruise. In rare cases, a blood draw can cause fainting. If you have fainted before when your blood was drawn please let the person drawing your blood know. Only trained people will draw your blood.

# Bone marrow biopsy and bone marrow aspirate

Bone marrow aspirate and/or biopsy are each performed using a hollow needle to remove a small sample of bone marrow. Before the biopsy, a local anesthetic is used to numb the area where the needle(s) will be inserted. The sterile procedure may cause discomfort, pain, bleeding, scarring or infection at the site of the aspirate and/or biopsy.

#### **C4. REPRODUCTIVE RISKS**

# Risks to women who could become pregnant

The drugs in this project might affect a baby, before or after the baby is born. We do not know if the drugs cause(s) harm to a baby, so we do not want anyone who might be pregnant to enter the project. You should not become pregnant or nurse a baby while in this project. You must tell the research doctor right away if you think you are pregnant. You will be asked to have a pregnancy test to be sure you are not pregnant at the start of the project.

If you become pregnant during the project, you will be dropped from participation for safety reasons. If you become pregnant while you are taking this experimental drug we ask that you inform the research doctor immediately. The research doctor will ask you for written permission to obtain information from you or your obstetrician on your pregnancy and the health of the baby.

#### Risks of fathering a child

You should not father a baby while taking part in this project because it is unknown if the drugs could affect a baby. If your partner is able to become pregnant, one or both of you must use some form of effective birth control. You must tell the research doctor right away if you think your partner is pregnant.

If you think that you have fathered a baby while you are taking this experimental drug, we ask that you inform the research doctor immediately. At that time, the research doctor will ask permission of your partner for the use and disclosure of her health information regarding the pregnancy. She will be asked to sign a separate consent form. She can choose to do this or not. She will be asked to sign this form to allow your research doctor to contact her obstetrician to collect information on the progress of the pregnancy and its outcome. The research doctor will make this information available to the sponsor for safety monitoring.

# Birth control methods for all subjects

Check with the research doctor about the birth control methods needed for this project and how long to use them. Some methods might not be good enough for this project. If you are having sex that could lead to pregnancy, you should use birth control while you are in this project. This may include:


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

Not having vaginal sex (abstinence)

- Taking birth control pills orally
- Having birth control shots or patches such as Depo-Provera
- Surgical sterilization (hysterectomy or tubal ligation)
- Use of an intrauterine device (IUD)
- Use of diaphragm with contraceptive jelly
- Use of condoms with contraceptive foam
- Use of diaphragm with condoms ("double barrier")
- Limiting sexual activity to a male partner who has had a vasectomy

## C5. ARE THERE ANY BENEFITS TO TAKING PART IN THE PROJECT?

We don't know if this study will help you. Your condition may get better but it could stay the same or even get worse. We hope the information from this study will help us develop better treatments for acute GVHD.

# D1. ARE THERE ANY COSTS TO BEING IN THE PROJECT?

Most of the medical care that you will receive in this project is considered routine care for your condition and would be recommended whether or not you join the project. Costs for routine care will be billed to you or your insurance carrier.

Activities / costs that are part of the project will not be billed to you or your insurance company. These are the study drug, Tildrakizumab, research samples and the process and shipping of research samples. Some insurers will not pay for drugs, tests or hospitalization that are part of research, so check with your insurer before you join this project. If you have questions regarding costs, please contact Dr. Runaas.

If you participate in this research, the costs of any necessary emergency medical treatment in the event of a research-related injury will be billed to you or your health insurance.

### D2. WILL I BE PAID FOR PARTICIPATING IN THE PROJECT?

There is no payment for being in this project.

# D3. WHAT OTHER HEALTHCARE CHOICES DO I HAVE?

You do not have to join this project. You are free to say yes or no. If you do not join this project, your research doctor can discuss other healthcare choices with you.

Your other choices may include:

- Joining a different research project
- The procedure or drug offered to you may also be available without being in any research project.

The research doctor can explain both the possible benefits and the risks of other options that are available to you.


**Informed Consent for Research** 


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

### D4. WILL I BE GIVEN NEW INFORMATION ABOUT THE PROJECT?

If we learn any important new information about the drugs that might change your mind about being in the project, we will tell you about it right away. You can then decide if you want to stay in the project.

### D5. WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THE PROJECT?

Emergency medical treatment for injuries directly related to your participation in this research project will be provided to you. You or your health insurance will be billed for the costs of this emergency treatment. MCW will decide on a case by case basis if they will reimburse you or your insurer for emergency treatment costs. If your research-related injury requires medical care beyond this emergency treatment, you or your insurer will be responsible for the costs of this follow-up care.

At this time, there is no plan for any additional financial payments.

If you believe that you have been injured because of your participation in this project, contact the research doctors right away. Contact information: Dr. Runaas, 414-805-6700.

Nothing in this consent form affects any legal rights you may have nor does it release the investigator, the sponsor, the institution, or its agents from liability for negligence.

#### D6. WHO CAN ANSWER MY QUESTIONS ABOUT THE PROJECT?

- If you have more questions about this project at any time, you can call Dr. Runaas at 414-805-6700
- If you have questions about your rights as a research participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

# E. PERMISSION TO COLLECT, USE AND SHARE HEALTH INFORMATION

# E1. What health information will be collected and used for this project?

To be in this research project, the research team needs your permission to access, collect and use some of your health information. If you say no, you cannot be in the project. This information may come from questions we ask, forms we ask you to fill out, or your medical record, as described below. We will only collect and use information needed for the project.

The protected health information (PHI) originates from services you will or have received at one or more of the following locations: the Medical College of Wisconsin (MCW); BloodCenter of Wisconsin (BCW); Children's Hospital of Wisconsin (CHW); any Froedtert Health Affiliate-Froedtert Memorial Lutheran Hospital (FMLH), Inc.; Community Memorial Hospital (CMH) Menomonee Falls, Inc.; St. Joseph's Community Hospital (SJH) West Bend, Inc.; Froedtert & The Medical College of Wisconsin Community Physicians Clinics, Inc. (FMCWCP); the West Bend Surgery Center, LLC; and the Froedtert Surgery Center, LLC.


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# The health information to be collected and used for this project is:

- Hospital/Medical Records
- Physician/Clinical Records
- Lab and/or Pathology Reports
- Radiology Reports
- Biological Samples

# E2. Who will see the health information collected for this project?

The only MCW/Froedtert Hospital employees allowed to handle your health information are those on the research team, those on the Institutional Review Board (IRB) and those who check on the research activities to make sure the hospital's rules are followed.

If the costs of any necessary emergency medical treatment in the event of a research-related injury are billed to your health insurance, your health information may need to be disclosed to the insurer for billing purposes.

The research team may share your information with people who don't work at MCW/Froedtert Hospital because they planned, pay for, or work with us on this project. The federal Privacy Rule may no longer protect your health information once it leaves MCW/Froedtert Hospital. For this project, we plan to share information with those doctors, researchers or government representatives working with us on this project at the institutions or companies listed here:

- The U.S. Food and Drug Administration (FDA)
- Covance Laboratories and affiliates
- Sun Pharmaceutical Industries, Inc.
- Federal agencies such as the Department of Health and Human Services (the DHHS), the National Cancer Institutes / National Institutes of Health (the NCI/NIH) and the Office of Human Research Protections (the OHRP)
- Other regulatory agencies and/or their Designated Representatives
- Any independent ethics committee, which approved this study
- Those required by law

Because this project involves the use of drugs and/or devices, the FDA also has the right to inspect all project records.

We may record your research information, including results of tests and procedures done for research, in your Froedtert Hospital and/or Medical College of Wisconsin medical record. As a result, this research information may be seen by people allowed to see your medical records for healthcare operations or treatment, by those you allow to see your medical records by giving written permission, and by others when required by law.


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

We will not use your personal health information for a different project without your permission or the permission of a hospital research review board (IRB). Once all personal identification is removed from your health information, the information may be used for future research or distributed to another investigator for future research without additional informed consent from you or your legally authorized representative. The information might also be used or released for other purposes without asking you. Results of the project may be presented in public talks or written articles, but no information will be presented that identifies you.

# E3. What are the risks of sharing this health information?

One risk of taking part in a research project is that more people will handle your personal health information collected for this project. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the research doctor about whether this could apply to you.

# E4. How long will you keep the health information for this project?

If you sign this form, we plan to keep your information without any end-date in case we need to check it again for this project.

# E5. Can I cancel my permission to share this health information?

If you change your mind later and do not want us to collect or share your health information, you need to send a letter to:

Lyndsey Runaas, MD
Froedtert & the Medical College of Wisconsin
Division of Hematology and Oncology
9200 W. Wisconsin Avenue
Milwaukee WI 53226

The letter must say that you have changed your mind and do not want the researcher to collect and share your health information. At that time, we may decide that you cannot continue to be part of the project. We may still use the information we have already collected.

# F1. FOR MORE INFORMATION ABOUT THE PROJECT

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can look up this project by referring to the ClinicalTrials.gov number NCT04112810 or by asking the research team for a printed copy.


IRB Protocol Number: 35737

IRB Approval Period: 12/13/2022 - 8/14/2023

**EFFECTIVE** 

December 13, 2022

MCW/FH IRB

# **CONSENT TO PARTICIPATE**

# By signing my name below, I confirm the following:

- I have read (or had read to me) this entire consent document.
   All of my questions have been answered to my satisfaction.
- The project's purpose, procedures, risks and possible benefits have been explained to me.
- I agree to let the research team use and share the health information and other information gathered for this project.
- I voluntarily agree to participate in this research project. I agree to follow the procedures as directed. I have been told that I can stop at any time.

**IMPORTANT:** You will receive a signed and dated copy of this consent form. Please keep it where you can find it easily. It will help you remember what we discussed today.

| Subject's Name please print | Subject's Signature | Date |
|---|---|---|
| Name of Witness (if applicable) please print (for short form consent process, or consent of blind or illiterate subject) | Signature of Witness | Date |
| Rationale for Use of Witness | | |
| ☐ Subject has limited/no literacy | ☐ Sponsor requirement | |
| ☐ Subject has limited English | Other | |
| proficiency | | |
| ☐ Subject has limited/no vision | | |
| * Name of person discussing/<br>obtaining consent please print | Signature of person discussing/obtaining consent | Date |
| * A manufact of the wassers to any tweire | ad and authorized by the Dringinal Invi | antimator to not an |

\* A member of the research team trained and authorized by the Principal Investigator to act on her/his behalf in obtaining informed consent according to the protocol. The Principal Investigator is responsible and accountable for the research project.

